CLINICAL TRIAL: NCT00581529
Title: Partial Breast Irradiation Using Accelerated Intensity Modulated Radiotherapy in Early Stage Breast Cancer After Breast-Conserving Surgery
Brief Title: Partial Breast Irradiation Using Accelerated Intensity Modulated Radiotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The trial was terminated early because fair/poor cosmesis developed in 7 of 32 women.
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCC 2004.020; IRB #2004-0459 & HUM 44980 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2007-12-20; First posted 2007-12-27 (Estimated); Results first posted 2014-08-28 (Estimated); Last update posted 2017-10-31 (Actual); Status verified 2017-09

CONDITIONS: Breast Cancer
Keywords: breast
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Radiotherapy (Experimental): IMRT (Intensity-modulated Radiation Therapy), 3.85 Gy per fraction, bid, for 5 consecutive days for a total dose of 38.5 Gy.
  Interventions: Radiation: IMRT

INTERVENTIONS:
Radiation: IMRT — Patients on protocol will be treated with accelerated radiotherapy, 3.85 Gy per fraction, bid, for 5 consecutive days for a total dose of 38.5 Gy.

SUMMARY:
This is a phase I- II feasibility study for delivering partial breast irradiation (PBI) in selected patients with early stage, lymph node negative, breast cancer after breast-conserving surgery using accelerated Intensity Modulated Radiotherapy (IMRT).

DETAILED DESCRIPTION:
This is a non-randomized Phase I-II feasibility study of partial breast irradiation with accelerated IMRT technique. In this study, patients will be eligible if the estimated risk of breast cancer elsewhere in the breast (beyond the tumor bed) is low. The radiation treatment will be available to women who are older than 40 years, have a DCIS (Ductal carcinoma in situ) or T1, N0, M0, (AJCC classification, version 6.0), non-lobular infiltrating carcinoma treated with breast-conserving surgery.

Patients will undergo a pre-treatment planning free breathing CT with 5mm cuts in the treatment position, on a breast board, with both arms extended above their head that will be used to plan the traditional two field (tangent) plan. An Active Breathing Control (ABC) device will be used to minimize target motion due to breathing during a second CT scan. The lumpectomy cavity will be identified and delineated, and margins of approximately 1.5 cm in three dimensions will be used to allow for subclinical tumor extension and daily set-up error. The organs at risk (heart, lungs, contralateral breast) will be contoured on both CT scans. An inverse planning system and optimization tools will be employed in order to achieve the best IMRT plan (to minimize the dose to the heart, lungs and contralateral breast), that will be compared to the two field plan. If the IMRT plan is shown to be the optimal one, in terms of doses to organs at risk, then the patient will be enrolled in the protocol and will proceed with the treatment. Treatment will start approximately two weeks after the planning CT is obtained. All patients on protocol will be treated with accelerated radiotherapy, 3.85 Gy per fraction, bid, for 5 consecutive days for a total dose of 38.5 Gy.

ELIGIBILITY:
Inclusion Criteria:

* Patient with unifocal histologically proven breast cancer, with or without calcifications in mammogram.
* DCIS (Ductal carcinoma in situ) (Tis, Stage 0)
* Non-lobular infiltrating carcinoma, maximum of 2 cm in diameter. (T1, Stage I)
* The patient was operated on and the tumor was excised with lumpectomy
* The tumor is reported with negative margins >3 mm, as per our hospital protocol.
* For invasive carcinoma, axillary lymph nodes are negative by sentinel lymph node (SLN) mapping and biopsy or by formal axillary lymph node dissection.
* The patient is over 40 years old with life expectancy of at least 5 years
* Karnofsky status must be at least 70. See appendix I.
* Pre- and post-menopausal women are eligible for entry.
* The patient must be aware of the neoplastic nature of her disease and must be willing to consent after being informed of the potential benefits, side effects and risks of radiotherapy. Institutional Review Board approval of this protocol and a consent form is required.

Exclusion Criteria:

* No concurrent or neoadjuvant chemotherapy is allowed. Patient is permitted to be treated with chemotherapy or hormone therapy only after completion of the radiation treatment.
* Patients with diffuse calcifications, multifocal or multicentric disease, lymph-vascular invasion are excluded.
* Patients cannot participate if there is extensive LCIS (Lobular carcinoma in situ) in specimen or extensive DCIS.
* Patients are excluded if systemic disease is present or the patient has been irradiated to the ipsilateral breast or the chest wall.
* Patients who are carriers of BRCA 1/2 mutations or at high risk for hereditary breast cancer due to strong family history (more than one pre-menopausal family member with breast cancer or any ovarian cancer) are excluded because of the increased potential for in-breast recurrence elsewhere in the breast in the absence of whole breast radiotherapy.
* Patients with scleroderma, or systemic or discoid lupus are excluded due to the potential for significant radiotherapy associated toxicity.
* Pregnant woman cannot participate in the study.
* Patients who have serious medical problems which would limit survival to <5 years or a psychiatric condition which would prevent informed consent cannot participate.
* Patients who are unable to lie on their back and raise their arms above their heads in the treatment planning position for radiotherapy are excluded.
* Patients that have mammographically occult disease are excluded.

Min Age: 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2004-11; Primary Completion 2010-10 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori J Pierce, MD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Radiotherapy: Patients on protocol will be treated with accelerated radiotherapy, 3.85 Gy per fraction, bid, for 5 consecutive days for a total dose of 38.5 Gy.
Period: Overall Study
Arm/Group | Radiotherapy
Started | 34
Completed | 34
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 34 for patients were enrolled and treated. 2 patients were excluded from all analysis due to fair baseline cosmesis. 2 additional patients underweant mastectomies and were therefore excluded from analysis (comsesis could not be assessed at 5 years). 30 patients were analyzed.
Arm/Group | Radiotherapy
Number analyzed (Participants) | 30
Age, Continuous [Median (Full Range); unit: years] | 56 [40 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30
  Male | 0
Laterality [Number; unit: participants] — Left or right breast
  participants
    Left Breast | 9
    Right Breast | 21
Histology [Number; unit: participants] — Breast cancer histology: Ductal carcinoma in situ (DCIS) or Invasive ductal carcinoma (IDC).
  participants
    DCIS | 16
    IDC | 14
Chemotherapy [Number; unit: participants] — Did participant receive chemotherapy following APBI (Accelerated partial breast irradiation)?
  participants
    Yes | 5
    No | 25
Endocrine Therapy [Number; unit: participants] — Did participant receive endocrine therapy following APBI (Accelerated partial breast irradiation)?
  participants
    Yes | 19
    No | 11
Re-excision [Number; unit: participants] — Did patients required a second surgical excision to achieve final negative margins?
  participants
    Yes | 15
    No | 15

OUTCOME MEASURES:

1. Primary Outcome: Rate of Local Control at 5 Years
Description: The primary objective was to determine the rate of local control (the arrest of cancer growth at the site of origin) of cancer in the treated breast at 5 years following breast-conserving surgery and partial breast radiotherapy using IMRT.
Time Frame: 5 years
Population: 34 for patients were enrolled and treated.
Measure: Number; unit: percentage of participants
Groups:
- Radiotherapy: Accelerated radiotherapy, 3.85 Gy per fraction, bid, for 5 consecutive days for a total dose of 38.5 Gy.
  IMRT: Patients on protocol will be treated with accelerated radiotherapy, 3.85 Gy per fraction, bid, for 5 consecutive days for a total dose of 38.5 Gy.
Arm/Group | Radiotherapy
Number analyzed (Participants) | 34
percentage of participants | 97

2. Primary Outcome: Percentage of Participants That Experience Cosmetic Adverse Events (AEs)
Description: The primary outcome was to determine the rate of acute cosmetic adverse events and late cosmetic adverse events at follow-up visits over 5 years. To determine the rate of adverse events, the percentage of participants experiencing no cosmetic AEs, at least 1 grade 1 toxicity, at least 1 grade 2 toxicity, and at least 1 grade 3 toxicity were calculated.
Time Frame: 5 years
Population: 34 for patients were enrolled and treated. 2 patients were excluded from all analysis due to fair baseline cosmesis. 2 additional patients underwent mastectomies and were therefore excluded from analysis (cosmesis could not be assessed at 5 years). 30 patients were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Radiotherapy
Number analyzed (Participants) | 30
percentage of participants
  Experiences no toxicities | 23.3
  Experienced at least 1 grade 1 toxicity | 40
  Experienced at least 1 grade 2 toxicity | 30
  Experienced at least 1 grade 3 toxicity | 6.7

3. Secondary Outcome: Dosimetric and Volumetric Differences Between Treatment Plans for Partial Breast Irradiation and Other Treatment Planning Methods
Description: Dosimetric and volumetric differences between treatment plans for partial breast irradiation and other treatment planning methods for the target (partial breast) and organs at risk (e.g. heart, ipsilateral lung, contralateral breast)a subset of 20.
Time Frame: not specific
Population: At the time the study was written, we planned to compare treatment methods. Over the course of the study, it was determined additional analysis was not needed due to the analysis and publication of this outcome by several other investigators.
Arm/Group | Radiotherapy
Number analyzed (Participants) | 0

4. Secondary Outcome: Mean Percentage of Reference Volume Receiving 19.25 Gy and 38.5Gy for Patients With Acceptable and Unacceptable Cosmesis
Description: One of the studies secondary outcomes was to evaluate the impact of short term accelerated partial breast radiation therapy on cosmetic results. To determine the association between dosimetric factors and cosmesis, the mean percentage of prescription dose received to WBV (Whole breast volume: corresponding region typically encompassed by traditional tangent fields) was compared among participants who developed fair/poor (F/P) cosmetic outcomes (unacceptable cosmesis) and participants who maintained excellent/good (E/G) cosmetic outcomes (acceptable cosmesis).
Time Frame: 5 years
Population: 34 for patients were enrolled and treated. 2 patients were excluded from all analysis due to fair baseline cosmesis.
Measure: Mean (Full Range); unit: Percentage of reference volume
Arm/Group | Radiotherapy
Number analyzed (Participants) | 32
Percentage of reference volume
  Mean % receiving 19.25, Acceptable Cosmesis | 34.6 [16.6 to 49.2]
  Mean % receiving 19.25, Unacceptable Cosmesis | 46.1 [31.3 to 64.5]
  Mean % receiving 38.5, Acceptable Cosmesis | 15.5 [6.8 to 25.4]
  Mean % receiving 38.5, Unacceptable Cosmesis | 23.0 [14.0 to 29.5]

ADVERSE EVENTS:
Arm/Group | Radiotherapy
Serious Adverse Events (participants affected / at risk) | 8/34
Other Adverse Events (participants affected / at risk) | 34/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy (N=34)
Fever with Neutropenia (General disorders) | 2
Headache (Nervous system disorders) | 1
Fever (General disorders) | 1
Breast Volume/Hypoplasia (Reproductive system and breast disorders) | 1
Gastrointestinal Bleeding (Gastrointestinal disorders) | 1 — Patient has history of Crohn's Disease
Telangiectasia (Vascular disorders) | 1
Chest Pain (Cardiac disorders) | 1
Diverticulitis (Gastrointestinal disorders) | 1 — Patient has history of Crohn's Disease
Acute Myeloid Leukemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 — Due to treatment with Adriamycin.
Kidney Stones (Renal and urinary disorders) | 1
Aortic Aneurysm (Cardiac disorders) | 1 — Patient had history of aortic aneurysms.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Radiotherapy (N=34)
Pain (General disorders) | 8
Nipple/Areolar Deformity (Reproductive system and breast disorders) | 26
Breast Hypoplasia (Reproductive system and breast disorders) | 30
Breast Induration Fibrosis (Reproductive system and breast disorders) | 25
Telangeictasia (Reproductive system and breast disorders) | 7
Edema-Limb (General disorders) | 2
Fatigue (General disorders) | 17
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 20
Dry Skin (Skin and subcutaneous tissue disorders) | 11
Rash (Skin and subcutaneous tissue disorders) | 8
Burn (Skin and subcutaneous tissue disorders) | 2
Fibrosis/Deep Tissue (Skin and subcutaneous tissue disorders) | 3
Hypopigmentation (Skin and subcutaneous tissue disorders) | 3
Pruitis/Itching (Skin and subcutaneous tissue disorders) | 4
Anorexia (Metabolism and nutrition disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Wound Complication (Injury, poisoning and procedural complications) | 1
Skin Atrophy (Skin and subcutaneous tissue disorders) | 1
Congestive Heart Failure (Cardiac disorders) | 1
Secondary Malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

LIMITATIONS AND CAVEATS:
The trial was terminated early because fair/poor cosmesis developed in 7 of 32 women.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes